CLINICAL TRIAL: NCT04085679
Title: Implementation of a Strategy to Prevent Hospital Admission in Nursing Home Residents: Protocol of a Quasi-experimental Study
Brief Title: Multidisciplinary Mobile Unit for Preventing Hospitalization of Nursing Home Residents
Acronym: MMU-1
Status: Terminated | Type: Observational
Why Stopped: The local Healthcare authorities extended the planned intervention to all nursing homes of the district after the emergence of multiple outbreaks of severe COVID-19 in several nursing homes.
Sponsor: Azienda Ospedaliero-Universitaria di Parma (Other)
Responsible Party: Principal Investigator, Tiziana Meschi, Head of Geriatric-Rehabilitation Department, Azienda Ospedaliero-Universitaria di Parma
Other Study IDs: MMU-1
Record Dates: First submitted 2019-09-09; First posted 2019-09-11 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Frailty; Disability; Multimorbidity; Respiratory Failure; Abdominal Pain; Infection
Keywords: Multidisciplinary care; Hospital-community care integration; Mobile specialist team; Personalization of care; Nursing home
MeSH Terms: conditions — Frailty; Respiratory Insufficiency; Abdominal Pain; Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MMU active group: Subjects residing in nursing homes where the MMU care model has already been implemented
  Interventions: Other: Multidisciplinary Mobile Unit (MMU)
- MMU control group: Subjects residing in nursing homes where the MMU care model has not yet been implemented (ED visits performed in case of urgent clinical situations)

INTERVENTIONS:
Other: Multidisciplinary Mobile Unit (MMU) — MMU is called in case of urgent clinical situations involving patients residing in nursing home
  Groups: MMU active group

SUMMARY:
Elderly patients residing in nursing homes are particularly at risk of experiencing urgent medical problems needing admission to the Emergency Department (ED). This circumstance contributes to ED overcrowding, increases the risk of ward admission of elderly patients, and puts them at an even higher risk of hospitalization-related adverse events. The study hypothesis is that a complex intervention, delivered directly in nursing homes by hospital physicians in case of urgent medical problems, would contribute to reduce hospitalization of older nursing home residents.

The intervention consists in a hospital-based "multidisciplinary mobile unit" (MMU), composed of a hospital specialist and a resident in emergency-urgency medicine who are coordinated by a senior physician serving as "flow manager". The team is active on work days, 8 am to 6 pm, and is activated by general practitioners of nursing homes, in case of urgent medical needs of one of the residents. The activation is made by a phone call to the "flow manager", who triages the clinical needs of the case. The output of the phone consultation may include therapeutic advice provided by phone, immediate on-site visit by the MMU team (specialist and resident), scheduled visit by the MMU team, or direct admission to the hospital unit where MMU is based, avoiding ED visits. The MMU team is provided with a portable ultrasound system, an essential set of drugs and medical devices useful in a urgency setting (central venous lines, nasogastric tubes, rectal tubes, bladder catheters). During on-site visits, the MMU team performs diagnosis, stabilization and therapeutic advice, with the mission of avoiding ED visits and hospital admissions whenever possible.

The MMU intervention is already active in two nursing homes, since December 2018. The aim of this prospective, pragmatic, multicenter, quasi-experimental study (sequential design with two cohorts) is to test the effects of the implementation of the MMU care model in terms of reduction of unplanned hospitalization rates (primary outcomes), mortality, health service use and costs (secondary outcomes).

Two nursing homes (i.e., the ones who already benefit from the intervention) will serve as study group, and two nursing homes with similar geographical location will serve as control group. All residents of the participating nursing homes will be eligible for study inclusion. The study will last for 18 months, and a number of 338 residents is planned for inclusion.

DETAILED DESCRIPTION:
The study is based in the University Hospital of Parma, which has a catchment area of more than 400,000 inhabitants, of whom 22.3% is over 65 years old. It provides the only Emergency service of the district, and it ranks fourth in Italy by number of ED visits (yearly average of over 110,000). The average admission rate of the adult ED population is 18%, of which 65% concern people older than 65.

In the last two decades, the University Hospital of Parma has implemented several innovative initiatives to manage the hospital flow of frail multimorbid patients and their complex needs. These initiatives included bed management to avoid "bed-blockers", physician accountability for the discharge process, and creation of a dedicated hospital unit, organized by intensity of care to anticipate the needs of these patients preserving high performance indices. This unit, called Internal Medicine and Critical Subacute Care Unit, performs over 3,500 urgent admissions of frail multimorbid elderly patients per year, with an average length of stay that in 30% of cases is lower than 3 days.

Participating nursing homes are public facilities which ensure the presence of nursing staff 24 hours a day and of a physician at least 4 hours a day (high-intensity care facilities). The possible role of distance to the hospital is considered by including in each group one nursing home located next to the hospital and one located >5 km of distance.

This study follows a multimethod approach, based on the MRC framework for developing and evaluating complex interventions, including the development, feasibility assessment, and evaluation phases.

1. Development of the intervention First, the different types of approaches reported in the literature, described above, were considered. The "prevention approach", interventions conducted in nursing homes, was chosen as the most suitable strategy to integrate the hospital's organizational model already in place, as it can target both hospitalization rates and ED overcrowding, allowing to intervene before the person accesses the hospital.

   Available evidence also prompted us to opt for a multicomponent approach. In fact, data from qualitative interviews reveal that the decision to transfer residents to hospital may be influenced by different factors, such as staffing and skill mix in the nursing homes, treatment options available in the facility, end-of-life decision-making, and communication and bureaucratic requirements. This multifactorial association means that a multicomponent intervention is likely to be more effective than a single-component intervention.

   The choice of employing a mobile geriatric specialist service was supported by the positive results obtained by the two controlled studies which examined similar interventions. One study evaluated a service where a physician did regular and on-call visits intended to provide services otherwise associated with hospitalization. The other study evaluated an ambulant team with a nurse and a physician, doing comprehensive geriatric assessments of residents as well as reviewing medications and providing support to staff. The proposed intervention does not involve a nurse, unlike the second of the mentioned studies, because in the participating facilities nursing staff is available 24 hours a day. Unlike the experience of the second study, moreover, periodic visits on site will not be performed in the present investigation, since routine clinical management and scheduled follow-up is already performed by nursing home physicians.

   Finally, medical hospital staff was preferred to community geriatricians, on the assumption that older patients may feel more comfortable being handled by physicians who may have already cared for them at the hospital. Moreover, hospital staff enables direct patient referral to the ward. Finally, this allows the use of diagnostic technologies available at the hospital, which can be used immediately without the need for hospital admission.

   The MMU care model intervention The model hinges on the strong collaboration between hospital and nursing home staff to provide residents with patient-centered care. It entails a multicomponent intervention which is integrated in standard care and comprises three steps: 1) MMU team activation, 2) on site visit by a team of physicians with geriatric expertise, 3) interdisciplinary care planning.

   Step 1: MMU team activation

   Patient selection is necessary to ensure that available resources are used for patients who may really benefit. To this end, the nursing home physician contacts by phone the "flow manager", a skilled internist with strong clinical expertise, organizational attitude and managerial training, during the 8 a.m.-6 p.m. time frame, Monday to Friday. The phone consultation is reported on a form containing the description of the patient's clinical condition and a summary of the conversation. The form also indicates which decision was reached among the following 6 not mutually exclusive options:
   1. The patient can be managed by nursing home staff, therapeutic advice is provided by phone
   2. Remote reassessment is scheduled after a number of hours agreed upon by the team
   3. The MMU team is dispatched for evaluation, treatment and stabilization on site
   4. A significant change in vital parameters is observed which requires immediate activation of emergency services
   5. Direct hospital admission is considered necessary
   6. Ambulatory outpatient visits or tests are planned

   Step 2: on site visit by a team of physicians with geriatric expertise Visits at the nursing home are performed by two members of the MMU team: an expert hospital physician chosen on a case-by-case basis among the clinical staff of the Internal Medicine and Critical Subacute Care Unit, which comprises internists, gastroenterologists, geriatricians, specialists in clinical nutrition, depending on the disease or clinical problem that must be treated, and a specifically trained resident in Emergency Medicine.

   The team is provided with a car to reach the nursing homes, a portable ultrasound system, and an essential set of drugs and medical devices useful in an emergency setting. The ultrasound system is equipped with three probes (convex, linear, and phased-array) for performing thoraco-pulmonary, cardiac, vascular, abdominal and soft tissue ultrasound, when required. Available drugs include those that can be administered intravenously for treating urgent conditions (e.g. loop diuretics, steroids, fluids, antibiotics). Devices include central and peripheral venous lines, naso-gastric and rectal tubes and bladder catheters. Blood tests can also be performed.

   Step 3: interdisciplinary care planning. Based on the results of the visit and of any performed investigations, the MMU team formulates personalized advice and referrals, and discusses these with the nursing home physician. If stabilization on site is not deemed possible, the MMU team plans a direct admission to the Internal Medicine and Critical Subacute Care Unit, thus avoiding ED access. The planning and the final outcome of the intervention are recorded in the second part of the form.
2. Feasibility assessment A pilot phase of 5 months (December 2018-April 2019) was conducted in two nursing homes in order to look at feasibility of the MMU care Model described above. Before the intervention was introduced, meetings were held with nursing home staff to agree on activation modalities.

   In this period, 99 phone calls were received, of which 84 required MMU team onsite visits, and 15 were managed with remote consultancy. Of the latter, 3 required direct admission after remote phone consultancy. Only 4 of the 84 patients visited onsite required direct admission. One patient was sent to the ED for massive intestinal bleeding.

   This phase demonstrated the feasibility of the intervention, and did not highlight any need for modifications.
3. Evaluation phase Aim and objectives The study aim is to verify the effects of the implementation of the MMU care model tested in the pilot phase.

Primary objective is to verify reduction of unplanned hospitalization rates in the nursing homes of the intervention group compared to the nursing homes in the control group. Secondary objectives are to measure the effects of the intervention in terms of mortality, health service use, and costs.

Study Design. This study is a prospective, pragmatic, multicenter, quasi-experimental study (sequential design with two cohorts), in which usual nursing home care is compared to care provided by applying the MMU model.

Study Population. All residents of the participating nursing homes are eligible, regardless of their clinical status. Residents who do not provide informed consent will be excluded.

Usual Care. Patients in the control cohort receive usual care, which means the actions to take are decided by the nursing home staff. Generally, this implies that patients who are clinically unstable, or require urgent instrumental tests, will be sent to the ED.

Measures. Baseline variables. Demographic data on gender and age are collected by chart review.

Outcome variables. The primary outcome is hospitalization rate, considering at the numerator all unplanned admissions occurred during a 1-year period, and at the denominator the sum of the person-time of the at risk population (days of stay at the nursing home). For the intervention group, the numerator corresponds to options c) and d) defined in "Step 1: MMU team activation".

Secondary outcomes:

* Crude all-cause Death Rate (CDR): the number of deaths during a 1-year period on person-time of the at risk population
* Hospital Mortality rate: the frequency of patients who die while in the hospital (death rate/1000)
* Length of stay (LOS): the duration of a single episode of hospitalization. Inpatient days are calculated by subtracting day of admission from day of discharge.
* Adverse events or complications: frequency of events occurred within 48 hours from MMU team activation and subsequent patient stabilization, for which hospital access becomes necessary.
* Costs analysis, comparing the cost differences in the two groups

Data Collection. Patient demographic and clinical characteristics are collected at baseline to describe the study population and determine factors associated with hospital rate. Participants' files and electronic data are stored securely at the study site (e.g. locked area, password protected hard- and software). Data integrity will be scrutinized with several strategies (e.g. valid values, range checks, consistency checks). Patient data are only identifiable with the unique participant's number. Personal information will be collected and saved in a separate file (on a different server) which can only be accessed by the Principal Investigator (PI). This information will be used by the PI to retrieve data on any hospital admissions (length of stay, in-hospital death …) from administrative databases (discharge summaries, ED data, Death Registry). Residents' identification data will be deleted once the study is completed, making the dataset anonymous. All study protocol authors will have access to the anonymous dataset.

Cost analysis. The investigators will identify the changes in net costs associated with one-year exposure to the intervention, consisting in the induced costs due to incremental resource inputs for carrying out the intervention and hospital health service utilization costs. Staffing costs will be calculated considering the time spent by the professionals involved in the intervention. Non-staff running costs include expenses of MMU staff travelling to and from the nursing home. The health service utilization costs will be identified based on the Diagnosis Related Group (DRG) system.

Statistical Methodology. Sample size calculation. The number of subjects to include was estimated using the findings of one study, a large quasi-experimental trial. Thus, considering 56 cases vs 32 cases per 100 residents, and using a 2-sided, large-samples z-test of the Poisson incidence rate difference at a significance level of 0.05, and with a power of 0.90, overall 338 residents should be enrolled.

Statistical analysis. Descriptive statistics will be used to summarize patient populations and will be presented as means and standard deviations (SD) when normally distributed, or as medians and interquartile ranges (IQR).

For the primary analysis the investigators will used Poisson regression with robust standard errors (SEs) to evaluate relative differences in hospital rates among the two cohorts while adjusting for demographic characteristics.

Concerning the secondary outcomes, the following analyses will be performed:

* Rates will be compared considering the quotient between the intervention and control groups
* A lognormal model will be used to compare in-hospital LOS.
* Chi square tests will be conducted for categorical data as adverse events or complications
* For costs, the investigators will use the following equations to summarize the annual net costs associated with the implementation of the intervention. Any costs with negative values mean "savings" and any costs with positive values mean "losses". Net costs ˆ A…(intervention costs) +‡ B (Costs for differences in hospital health service utilization) where: A= intervention: staffing costs+intervention: non- staff costs and B= Costs for differences in inpatient care utilization. Therefore, the net costs arising from one-year implementation of the intervention as compared with the current practice will be obtained, where a negative value of net costs represents "cost-saving" and a positive value represents "not cost-saving"

The demographic and clinical variables which influence the outcome with a p value<0.20 in the univariate analysis will be included in the Poisson regression model.

The analyses will be performed using SAS 8.2 (SAS Institute, Cary, NC, USA) and STATA-SE 11 (Stata Corp LP, College Station, TX, USA).

ELIGIBILITY:
Inclusion Criteria:

* All residents of the participating nursing homes, regardless of age, gender or clinical conditions

Exclusion Criteria:

* Unwillingness to sign informed consent form (patient him/herself or legal representatives)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All subjects residing in the nursing homes participating to the study will be eligible for inclusion, regardless of their clinical conditions. Participating nursing homes are public facilities which ensure the presence of nursing staff 24 hours a day and of a physician at least 4 hours a day (high-intensity care facilities). The possible role of distance to the hospital is considered by including in each group one nursing home located next to the hospital and one located >5 km of distance.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Hospitalization rate | 1 year
  Calculated as all unplanned admissions divided per the sum of the person-time of the at-risk population (days of stay at the nursing home)

SECONDARY OUTCOMES:
Crude all-cause death | 1 year
  Number of deaths on person-time of the at-risk population
Hospital mortality rate | 1 year
  The frequency of patients dead while in hospital (death rate/1000)
Length of hospital stay | 1 year
  Duration of a single episode of hospitalization, with inpatient days calculated by subtracting day of admission from day of discharge
Adverse events or complications | 1 year
  Frequency of events occurred within 48 hours from MMU team activation and subsequent patient stabilization, for which hospital access becomes necessary
Cost analysis | 1 year
  Hospitalization-related costs

CONTACTS AND LOCATIONS:
Overall Officials: Tiziana Meschi, M.D., Principal Investigator — Azienda Ospedaliero-Universitaria di Parma (Parma University Hospital)
Locations (1):
- UO Medicina Interna e Lungodegenza Critica, Azienda Ospedaliero-Universitaria di Parma, Parma, Emilia-Romagna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aminzadeh F, Dalziel WB. Older adults in the emergency department: a systematic review of patterns of use, adverse outcomes, and effectiveness of interventions. Ann Emerg Med. 2002 Mar;39(3):238-47. doi: 10.1067/mem.2002.121523. PMID 11867975
- [Background] Arendts G, Howard K. The interface between residential aged care and the emergency department: a systematic review. Age Ageing. 2010 May;39(3):306-12. doi: 10.1093/ageing/afq008. Epub 2010 Feb 22. PMID 20176712
- [Background] Buurman BM, Hoogerduijn JG, van Gemert EA, de Haan RJ, Schuurmans MJ, de Rooij SE. Clinical characteristics and outcomes of hospitalized older patients with distinct risk profiles for functional decline: a prospective cohort study. PLoS One. 2012;7(1):e29621. doi: 10.1371/journal.pone.0029621. Epub 2012 Jan 4. PMID 22238628
- [Background] Caminiti C, Meschi T, Braglia L, Diodati F, Iezzi E, Marcomini B, Nouvenne A, Palermo E, Prati B, Schianchi T, Borghi L. Reducing unnecessary hospital days to improve quality of care through physician accountability: a cluster randomised trial. BMC Health Serv Res. 2013 Jan 10;13:14. doi: 10.1186/1472-6963-13-14. PMID 23305251
- [Background] Corazza GR, Formagnana P, Lenti MV. Bringing complexity into clinical practice: An internistic approach. Eur J Intern Med. 2019 Mar;61:9-14. doi: 10.1016/j.ejim.2018.11.009. Epub 2018 Dec 6. PMID 30528261
- [Background] Craig P, Dieppe P, Macintyre S, Michie S, Nazareth I, Petticrew M; Medical Research Council Guidance. Developing and evaluating complex interventions: the new Medical Research Council guidance. BMJ. 2008 Sep 29;337:a1655. doi: 10.1136/bmj.a1655. PMID 18824488
- [Background] Diaz-Gegundez M, Paluzie G, Sanz-Ballester C, Boada-Mejorana M, Terre-Ohme S, Ruiz-Poza D. [Evaluation of an intervention program in nursing homes to reduce hospital attendance]. Rev Esp Geriatr Gerontol. 2011 Sep-Oct;46(5):261-4. doi: 10.1016/j.regg.2011.03.001. Epub 2011 Sep 23. Spanish. PMID 21944328
- [Background] Jay S, Whittaker P, Mcintosh J, Hadden N. Can consultant geriatrician led comprehensive geriatric assessment in the emergency department reduce hospital admission rates? A systematic review. Age Ageing. 2017 May 1;46(3):366-372. doi: 10.1093/ageing/afw231. PMID 27940568
- [Background] Limpawattana P, Phungoen P, Mitsungnern T, Laosuangkoon W, Tansangworn N. Atypical presentations of older adults at the emergency department and associated factors. Arch Gerontol Geriatr. 2016 Jan-Feb;62:97-102. doi: 10.1016/j.archger.2015.08.016. Epub 2015 Aug 21. PMID 26323650
- [Background] Mannucci PM, Nobili A, Pasina L; REPOSI Collaborators (REPOSI is the acronym of REgistro POliterapie SIMI, Societa Italiana di Medicina Interna). Polypharmacy in older people: lessons from 10 years of experience with the REPOSI register. Intern Emerg Med. 2018 Dec;13(8):1191-1200. doi: 10.1007/s11739-018-1941-8. Epub 2018 Aug 31. PMID 30171585
- [Background] Meschi T, Nouvenne A, Maggio M, Lauretani F, Borghi L. Bed-blockers: an 8 year experience of clinical management. Eur J Intern Med. 2012 Mar;23(2):e73-4. doi: 10.1016/j.ejim.2011.11.012. Epub 2011 Dec 6. No abstract available. PMID 22284263
- [Background] Meschi T, Ticinesi A, Prati B, Montali A, Ventura A, Nouvenne A, Borghi L. A novel organizational model to face the challenge of multimorbid elderly patients in an internal medicine setting: a case study from Parma Hospital, Italy. Intern Emerg Med. 2016 Aug;11(5):667-76. doi: 10.1007/s11739-016-1390-1. Epub 2016 Feb 4. PMID 26846233
- [Background] Roberts DC, McKay MP, Shaffer A. Increasing rates of emergency department visits for elderly patients in the United States, 1993 to 2003. Ann Emerg Med. 2008 Jun;51(6):769-74. doi: 10.1016/j.annemergmed.2007.09.011. Epub 2007 Dec 11. PMID 18069088
- [Background] Salvi F, Morichi V, Grilli A, Giorgi R, De Tommaso G, Dessi-Fulgheri P. The elderly in the emergency department: a critical review of problems and solutions. Intern Emerg Med. 2007 Dec;2(4):292-301. doi: 10.1007/s11739-007-0081-3. Epub 2007 Nov 28. PMID 18043874
- [Background] Samaras N, Chevalley T, Samaras D, Gold G. Older patients in the emergency department: a review. Ann Emerg Med. 2010 Sep;56(3):261-9. doi: 10.1016/j.annemergmed.2010.04.015. PMID 20619500
- [Background] Santosaputri E, Laver K, To T. Efficacy of interventions led by staff with geriatrics expertise in reducing hospitalisation in nursing home residents: A systematic review. Australas J Ageing. 2019 Mar;38(1):5-14. doi: 10.1111/ajag.12593. Epub 2018 Oct 7. PMID 30294903
- [Background] Schippinger W, Hartinger G, Hierzer A, Osprian I, Bohnstingl M, Pilgram EH. [Mobile geriatric consultant services for rest homes. Study of the effects of consultations by internal medicine specialists in the medical care of rest home residents]. Z Gerontol Geriatr. 2012 Dec;45(8):735-41. doi: 10.1007/s00391-012-0395-2. German. PMID 23184299
- [Background] Wyman JF, Hazzard WR. Preventing avoidable hospitalizations of nursing home residents: a multipronged approach to a perennial problem. J Am Geriatr Soc. 2010 Apr;58(4):760-1. doi: 10.1111/j.1532-5415.2010.02775.x. No abstract available. PMID 20398159
- [Derived] Nouvenne A, Caminiti C, Diodati F, Iezzi E, Prati B, Lucertini S, Schianchi P, Pascale F, Starcich B, Manotti P, Brianti E, Fabi M, Ticinesi A, Meschi T. Implementation of a strategy involving a multidisciplinary mobile unit team to prevent hospital admission in nursing home residents: protocol of a quasi-experimental study (MMU-1 study). BMJ Open. 2020 Feb 17;10(2):e034742. doi: 10.1136/bmjopen-2019-034742. PMID 32071189